CLINICAL TRIAL: NCT07029074
Title: Investigation of the Acute Effect of Inspiratory Muscle Training Applied at Different Intensities on Intercostal Muscle Oxygenation
Brief Title: Investigation of Inspiratory Muscle Training Applied at Different Intensities on Intercostal Muscle Oxygenation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Başak KAVALCI KOL, Principle Investigator, Kirsehir Ahi Evran Universitesi
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: AhiEvranU529
Record Dates: First submitted 2025-06-05; First posted 2025-06-19 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-06

CONDITIONS: Healthy
Keywords: muscle oxygenation; inspiratory muscle training; intercostal muscle
MeSH Terms: interventions — Maximal Respiratory Pressures

STUDY DESIGN:
Intervention Model Description: This study was designed as a single-blind randomized, placebo-controlled, crossover study.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sham inspiratory muscle training (Maximal inspiratory pressure (MIP) 0%) (Experimental): Individuals participating in the study will be randomly assigned sham inspiratory muscle training sessions maximal inspiratory pressure of 0% under the supervision of a specialist physiotherapist for 30 minutes.
  Interventions: Device: Sham inspiratory muscle training (MIP 0%)
- MIP 30% inspiratory muscle training (Experimental): Individuals participating in the study will be randomly assigned inspiratory muscle training sessions maximal inspiratory pressure of 30% under the supervision of a specialist physiotherapist for 30 minutes.
  Interventions: Device: MIP 30% inspiratory muscle training
- MIP 70% inspiratory muscle training (Experimental): Individuals participating in the study will be randomly assigned inspiratory muscle training sessions maximal inspiratory pressure of 70% under the supervision of a specialist physiotherapist for 30 minutes.
  Interventions: Other: MIP 70% inspiratory muscle training

INTERVENTIONS:
Device: Sham inspiratory muscle training (MIP 0%) — POWERbreathe Wellness (POWERbreathe International Ltd.., England, UK) device will be used for inspiratory muscle training.
  Arms: Sham inspiratory muscle training (Maximal inspiratory pressure (MIP) 0%)
Device: MIP 30% inspiratory muscle training — POWERbreathe Wellness (POWERbreathe International Ltd.., England, UK) device will be used for inspiratory muscle training.
  Arms: MIP 30% inspiratory muscle training
Other: MIP 70% inspiratory muscle training — POWERbreathe Wellness (POWERbreathe International Ltd.., England, UK) device will be used for inspiratory muscle training.
  Arms: MIP 70% inspiratory muscle training

SUMMARY:
In this study, it was aimed to investigate the acute effect of inspiratory muscle training of different intensities on intercostal muscle oxygenation in healthy individuals.

DETAILED DESCRIPTION:
The functional activity of the respiratory system must be regular and efficient in order to meet the oxygen needs of tissues and organs. The mechanical function of the respiratory system is significantly related to the working capacity of the respiratory muscles. The diaphragm is the primary muscle that provides respiratory functions among the respiratory muscles.The external intercostal muscles help with the inspiration, while the internal intercostal muscles help with the expiration. The basis of inspiratory muscle training is to reduce dyspnea, increase inspiratory muscle function and exercise tolerance. Inspiratory muscle training provides an increase in muscle strength by increasing inspiratory muscle strength, reducing metaboreflex activity and increasing blood flow to the muscles. Training is thought to minimize the effects of activation of inspiratory muscle metaboreflex in both healthy individuals and patients with heart failure. In chronic respiratory patients, forced inspiration effort reduces capillary perfusion of the respiratory muscles, thus increasing the oxygen demand of the muscle. Muscle oxygen saturation shows the oxygen uptake and oxygen consumption of the muscle. It aims to investigate the mechanisms involved in the metaboreflex response to respiratory fatigue in inspiratory muscle training, which severity will acutely reduce it more.

ELIGIBILITY:
Inclusion Criteria:

* Physically active (doing moderate intensity physical activity for at least 3 days a week for 150 minutes / week)
* Volunteer to participate in the study

Exclusion Criteria:

* Healthy individuals with any diagnosed chronic or systemic disease,
* Smoke 10 packs x years or more,
* Pneumonia or any acute infection,
* Psychiatric disorder will excluded in the study.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-07-23 (Actual); Primary Completion 2025-12-23 (Estimated); Study Completion 2026-06-23 (Estimated)

PRIMARY OUTCOMES:
Evaluation of intercostal muscle oxygenation | Second, Third and Fourth day
  Before the inspiratory muscle training sessions, the muscle oxygen saturation (SmO2) of the intercostal muscles in recovery during and after the training session will be measured using a Moxy® monitor (Moxy, Fortiori Design LLC, Minnesota, USA).
Evaluation of intercostal muscle total hemoglobin level | Second, Third and Fourth day
  Before the inspiratory muscle training sessions, total hemoglobin level (THb) of the intercostal muscles in recovery during and after the training session will be measured using a Moxy® monitor (Moxy, Fortiori Design LLC, Minnesota, USA).

SECONDARY OUTCOMES:
Evaluation of respiratory muscle strength | First day
  An electronic mouth pressure device will be used to evaluate respiratory muscle strength. Patients will have maximal inspiratory pressure and maximal expiratory pressure measured with a mouth pressure measuring device.
Evaluation of respiratory muscle endurance | First day
  The incremental threshold loading test will be used to evaluate respiratory muscle endurance. The PowerBreathe Wellness® (HaB International Ltd. Southam, UK) will be used in the incremental threshold loading test.
Evaluation of pulmonary function (Forced expiratory volume in the first second (FEV1)) | First day
  Measurement of FEV1 will be performed with spirometer according to the criteria of the American Thoracic Society and the European Respiratory Society.
Evaluation pulmonary function (Forced vital capacity (FVC)) | First day
  Measurement of FVC will be performed with spirometer according to the criteria of the American Thoracic Society and the European Respiratory Society.
Evaluation of pulmonary function (FEV1/FVC) | First day
  Measurement of FEV1/FVC will be performed with spirometer according to the criteria of the American Thoracic Society and the European Respiratory Society.
Evaluation of pulmonary function (Flow rate 25-75% of forced expiratory volume (FEF 25-75%)) | First day
  Measurement of FEF 25-75% will be performed with spirometer according to the criteria of the American Thoracic Society and the European Respiratory Society.
Pulmonary function (Peak expiratory flow (PEF)) | First day
  Measurement of PEF will be performed with spirometer according to the criteria of the American Thoracic Society and the European Respiratory Society.
Evaluation of physical activity level | First day
  The physical activity level of individuals will be evaluated using the short form of the International Physical Activity Questionnaire. A score is obtained by multiplying the metabolic equivalent (MET) value by days and minutes. When calculating the walking score, the walking time will be multiplied by 3.3 METs; when calculating the moderate intensity activity score, it will be multiplied by 4 METs; when calculating the vigorous activity score, it will be multiplied by 8 METs. Physical activity levels will be classified as physically inactive (3000 MET-min/week).

CONTACTS AND LOCATIONS:
Locations (1):
- Kırşehir Ahi Evran University, Physical Therapy and Rehabilitation Center, Cardiopulmonary Unit, Kırşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data will be stored in a locked cabinet.